CLINICAL TRIAL: NCT02666170
Title: Effects of 6 Months of Alpha-Lipoic Acid Treatment on Clinical, Endocrine ed Metabolic Features in Women Affected by PCOS
Brief Title: Effects of Alpha-acid Lipoic in PCOS Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Rosanna Apa, Professor, Catholic University of the Sacred Heart
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Alpha-Lipoic Acid 2016
Record Dates: First submitted 2016-01-21; First posted 2016-01-28 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Thioctic Acid

ARMS (1):
- therapy with alpha-lipoic acid daily for six months (Experimental)
  Interventions: Drug: Alpha-lipoic acid

INTERVENTIONS:
Drug: Alpha-lipoic acid

SUMMARY:
The aim of our study is to investigate the effects of six months treatment with alpha-lipoic acid on clinical, endocrine and metabolic features in women affected by PCOS. Menstrual pattern, anthropometric parameters, hirsutism score, ultrasound ovarian featureas, an oral glucose tolerance test and hormonal assays are evaluated before and after therapy.

ELIGIBILITY:
Inclusion Criteria:

* women with PCOS in accordance with Rotterdam criteria

Exclusion Criteria:

* pregnancy
* past history of cardiovascular diseases
* diabetes mellitus (or impaired glucose tolerance as determined by a standard 75 gr oral glucose tolerance test)
* hypertension
* significant liver or renal impairment
* other hormonal dysfunction (hypothalamic, pituitary, thiroidal or adrenal)
* neoplasms.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Number of cycles in six months of therapy | 6 months

SECONDARY OUTCOMES:
Hirsutism score | 6 months
  Ferriman-Gallwey score
Insulin levels | 6 months
androstenedione levels | 6 months
testosterone levels | 6 months
free androgen index | 6 months
total cholesterol | 6 months
LDL-cholesterol | 6 months
tryglycerides levels | 6 months
DHEAS levels | 6 months
AMH levels | 6 months